CLINICAL TRIAL: NCT06319131
Title: Comparative Effectiveness of Nadroparin Versus Transjugular Intrahepatic Portosystemic Shunt in Cirrhotic Patients With Refractory Asymptomatic Portal Vein Thrombosis：a Multicenter, Randomized Controlled Trial
Brief Title: Nadroparin Versus TIPS in Cirrhotic Patients With Refractory Asymptomatic PVT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai 6th People's Hospital (Other); ShuGuang Hospital (Other); Tongji Hospital (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tipharosis
Record Dates: First submitted 2024-03-11; First posted 2024-03-19 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Portal Vein Thrombosis
Keywords: portal vein thrombosis; liver cirrhosis; nadroparin; transjugular intrahepatic portosystemic shunt
MeSH Terms: conditions — Liver Cirrhosis | interventions — Portasystemic Shunt, Transjugular Intrahepatic; Nadroparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIPS group (Experimental): The cirrhotic patients with persistent PVT despite 6 months of anticoagulation therapy will receive transjugular-intrahepatic-portosystemic shunt.
  Interventions: Procedure: TIPS
- Nadroparin group (Active Comparator): The cirrhotic patients with persistent PVT despite 6 months of anticoagulation therapy will continue with the nadroparin therapy
  Interventions: Drug: Nadroparin

INTERVENTIONS:
Procedure: TIPS — Using the transjugular approach, TIPS was created under local anesthesia. The first branch of the left or right portal vein (PV) was punctured by RUPS-100 set guided by digital subtraction angiography. After successful access into PV, direct portography was performed and all visible varices and/or concurrent spontaneous portosystemic shunts (SPSS) were embolized with coils and n-butyl cyanoacrylate. A polytetrafluoroethylene-covered stent (Viatorr Endoprosthesis, GORE and Associates, Flagstaff, Arizona, USA) with a diameter of 8 mm was implanted and fully dilated.
  Arms: TIPS group
Drug: Nadroparin — Nadroparin calcium will be subcutaneously injected with the dose of 85IU/kg q12h
  Arms: Nadroparin group

SUMMARY:
The purpose of this study is to evaluate the comparative effectiveness of nadroparin versus transjugular intrahepatic portosystemic shunt in cirrhotic patients with refractory asymptomatic portal vein thrombosis using a design of a multicenter, randomized controlled trial

DETAILED DESCRIPTION:
This research project aims to investigate the efficacy and safety of anticoagulant therapy in patients with portal vein thrombosis (PVT) associated with liver cirrhosis. Building upon this, a randomized controlled study will be carried out for PVT patients with poor response to anticoagulant treatment. The study will compare the effects of transjugular intrahepatic portosystemic shunt (TIPS) and prolonged anticoagulant therapy. The ultimate goal is to provide high-quality clinical research evidence for interventional treatment of liver cirrhosis-associated PVT. This comprehensive approach aims to provide evidence-based medical guidance for optimizing the treatment pathway for refractory PVT in liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with liver cirrhosis
* Diagnosis of portal vein thrombosis through computed tomographic venography with a thrombus diameter exceeding 30% of the vessel diameter.
* Consent to participate in the clinical trial and the signing of an informed consent form.

Exclusion Criteria:

* Presence of acute symptoms such as fever, abdominal pain or bleeding, or of cavernous transformation
* Patients with Child-Pugh C.
* Pregnant or lactating women.
* With a history of liver cancer or other malignancy.
* Severe heart, lung diseases, or significant renal dysfunction.
* Allergies to anticoagulant medications, uncontrolled hypertension, history of cerebral hemorrhage, discovery of gastrointestinal ulcers, ulcerative colitis, subacute bacterial endocarditis, or other contraindications to anticoagulant drugs.
* On concomitant therapy of immunosuppressive drugs.
* With coagulation disorders other than liver disease.
* With active variceal bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
complete recanalization rate of PVT | 6 months
  Enhanced abdominal CT scan will be performed to assess the recanalization of PVT. The primary outcome is the complete recanalization.

SECONDARY OUTCOMES:
partial recanalization rate of PVT | 6 months
  Enhanced abdominal CT scan will be performed to assess the recanalization of PVT. Partial recanalization is defined as decrease of PVT more than 50%.
Bleeding rate | 6 months
  Bleeding events related to anticoagulant therapy. Bleeding events will be further classified into major and minor according to the established criteria outlined by the International Society of Thrombosis and Haemostasis
Mortality | 6 months
  Survival analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wang, MD, Principal Investigator — Shanghai Zhongshan Hospital

IPD SHARING:
Plan to Share IPD: Undecided